CLINICAL TRIAL: NCT04025736
Title: Intravenous Administration of Tranexamic Acid Significantly Improved Clarity of Visual Field in Arthroscopic Shoulder Surgery. A Prospective, Double-blind and Randomized Controlled Trial
Brief Title: Arthroscopic Shoulder Surgery With Administration of Intravenous Tranexamic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-BR-106-017
Record Dates: First submitted 2019-07-14; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Rotator Cuff Tears; Shoulder Arthorscopy Surgery; Surgical Blood Loss; Tranexamic Acid
Keywords: Tranexamic Acid; Shoulder Arthroscopy; Visual Clarity; Hemostasis
MeSH Terms: conditions — Rotator Cuff Injuries; Blood Loss, Surgical | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Inclusion criteria were Patients who were diagnosed with rotator cuff tear and failure of conservative treatment for more than 3 months. The tear size was measured by MRI and must be repairable. We excluded patients who did not provide permit, those had history of coagulopathy, who were under anticoagulation therapy before surgery, who had abnormal coagulation profile (prothrombin time or activated partial thromboplastin time) before surgery, who had renal or liver disorder, those who had uncontrolled hypertension (systolic pressure >180 mmHg), or who were allergy to local anesthetic agent or Tranexamic acid.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients received Tranexamic acid (Experimental): The patient was assigned as intervention group, TXA will be aspirated into a syringe. In TXA group, TXA 1000 mg (20 mL) was given intravenously 10 minutes before surgery.
  Interventions: Drug: Tranexamic Acid 100Mg/Ml Inj Vil 10Ml
- Patients received same volume of saline (Placebo Comparator): In the control group, the patient received 20ml saline intravenous also 10 min before surgery.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Tranexamic Acid 100Mg/Ml Inj Vil 10Ml — Tranexamic acid (TXA) is a synthetic analog of the amino acid lysine which acts by competitively blocking the plasminogen lysine-binding site and inhibiting fibrinolysis. Several studies showed that TXA could reduce both blood loss and the amount of blood transfusion after shoulder arthroplasty surgeries.
  Arms: Patients received Tranexamic acid
Drug: 0.9% Sodium Chloride Injection — Normal saline is a mixture of sodium chloride in water and has a number of uses in medicine. We use the same volume of normal saline as placebo.
  Arms: Patients received same volume of saline

SUMMARY:
Purpose: The study aimed to determine whether intravenous administration of tanexamic acid (TXA) before shoulder arthroscopic rotator cuff repair surgery can improve arthroscopy visual clarity. Methods: This is a prospective, double-blinded, randomized and placebo-controlled study. From May 2016 to April 2018, patients requiring arthroscopic rotator cuff repair were enrolled and randomly assigned to either the TXA group that received 1000mg tranexamic acid intravenously 10 minutes before surgery or the placebo group that received the same volume of plain saline. Patients with pre-existing liver/renal disease, coagulopathy, or concurrent use of anti-coagulation medications were excluded. The visual clarity was rated by a numeric rating scale from grade

1(poor) to grade 3(clear) every 15 minutes throughout the surgery. Secondary outcomes included estimated perioperative blood loss, operative time, degree of shoulder swelling, postoperative subjective pain score, inpatient duration and associated comorbidities were recorded. Both parametric and nonparametric methods were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with rotator cuff tear and failure of conservative treatment for more than 3 months. The tear size was measured by MRI and must be repairable.

Exclusion Criteria:

* Acute traumatic rotator cuff tear.
* History of coagulopathy
* Under anticoagulation therapy before surgery
* Abnormal coagulation profile (prothrombin time or activated partial thromboplastin time) before surgery
* Renal or liver disorder
* Uncontrolled hypertension (baseline systolic pressure >180 mmHg)
* Allergy to local anesthetic agent or TXA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Visual clarity during shoulder arthroscopic surgery. | Measure the percentage of grade 3 visual clarity after surgery through study completion, an average of 1 year.
  We use 3-grades visual clarity. grade 1 means poor visual clarity; 2 means fair clarity and 3 means good clarity. The visual clarity was scored in every 15 minutes during the operation scoring system to evaluate visual clarity during arthroscopic surgery. 4 Grade 1 means poor visibility (active bleeding that the vision was too poor to perform the operation); Grade 2 means fair visibility (minor bleeding that can interfere vision but surgery can still perform); Grade 3 means good visibility (clear vision without obvious blood).
Visual clarity during shoulder arthroscopic surgery. | Measure the whole surgery's mean visual clarity grade after surgery through study completion, an average of 1 year.
  We use 3-grades visual clarity. grade 1 means poor visual clarity; 2 means fair clarity and 3 means good clarity. The visual clarity was scored in every 15 minutes during

SECONDARY OUTCOMES:
patients' visual analog scale (VAS ) pain score on postoperative day 1 | measure on post operative day one's morning through study completion, an average of 1 year.
  The visual analog scale(VAS) for pain is a continuous scale comprised of a horizontal line, which was 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme (from 0 cm means no pain to 10cm means worst pain possible) for patients self-assessment of pain.
post operation shoulder swelling | measure on post operative day one's morning through study completion, an average of 1 year.
  (compared the circumference of shoulder post op day 1 to the day of admission which were measured at two sites: axillary and deltoid),
change of serum hemoglobin before and after operation | measure on post operative day one's morning through study completion, an average of 1 year.
  use the change of Hb to calculate estimate blood loss by Gross formula.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] van Montfoort DO, van Kampen PM, Huijsmans PE. Epinephrine Diluted Saline-Irrigation Fluid in Arthroscopic Shoulder Surgery: A Significant Improvement of Clarity of Visual Field and Shortening of Total Operation Time. A Randomized Controlled Trial. Arthroscopy. 2016 Mar;32(3):436-44. doi: 10.1016/j.arthro.2015.08.027. PMID 26524933
- [Result] Karaaslan F, Karaoglu S, Yurdakul E. Reducing Intra-articular Hemarthrosis After Arthroscopic Anterior Cruciate Ligament Reconstruction by the Administration of Intravenous Tranexamic Acid: A Prospective, Randomized Controlled Trial. Am J Sports Med. 2015 Nov;43(11):2720-6. doi: 10.1177/0363546515599629. Epub 2015 Sep 2. PMID 26337246
- [Result] Felli L, Revello S, Burastero G, Gatto P, Carletti A, Formica M, Alessio-Mazzola M. Single Intravenous Administration of Tranexamic Acid in Anterior Cruciate Ligament Reconstruction to Reduce Postoperative Hemarthrosis and Increase Functional Outcomes in the Early Phase of Postoperative Rehabilitation: A Randomized Controlled Trial. Arthroscopy. 2019 Jan;35(1):149-157. doi: 10.1016/j.arthro.2018.07.050. PMID 30611343
- [Result] Kirsch JM, Bedi A, Horner N, Wiater JM, Pauzenberger L, Koueiter DM, Miller BS, Bhandari M, Khan M. Tranexamic Acid in Shoulder Arthroplasty: A Systematic Review and Meta-Analysis. JBJS Rev. 2017 Sep;5(9):e3. doi: 10.2106/JBJS.RVW.17.00021. PMID 28902659